CLINICAL TRIAL: NCT04553016
Title: A Phase 1 Trial of ChAdOx1- and MVA-vectored Conserved Mosaic HIV-1 Vaccines in Healthy, Adult HIV-1-negative Volunteers in Eastern and Southern Africa.
Brief Title: A Study to Test Three Experimental HIV Vaccines in Healthy Adults.
Acronym: HIV-CORE 006
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University of Nairobi (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); London School of Hygiene and Tropical Medicine (Other); International AIDS Vaccine Initiative (Network); Imperial College London (Other); Center for Family Health Research in Zambia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HIV-CORE 006
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: HIV-1-infection
Keywords: HIV; vaccine; adenovirus; poxvirus; ChAdOx1; MVA
MeSH Terms: conditions — Adenoviridae Infections | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain blinding, all volunteers will receive two injections with half dose into the deltoid region of each arm of ChAdOx1.tHIVconsv1 or placebo at enrolment, and two injections (MVA.tHIVconsv3 or placebo into one deltoid region and MVA.tHIVconsv4 or placebo into the other) at 4 weeks after enrolment.
  Unblinded study pharmacist(s) staff at each site will be responsible for investigational medicinal product preparation and accountability. All other site staff and all trial volunteers will be blinded to treatment assignment (i.e., active versus placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: Vaccine (Experimental): At Week 0, volunteers receive 5.0 x 10^10 virus particles (vp) of ChAdOx1.tHIVconsv1 (C1) administered intramuscularly (IM). The dose is divided in 2 and administered in the deltoid muscle of each arm.
  At week 4,1.0 x 10^8 Plaque forming units (PFU) of MVA.tHIVconsv3 (M3) administered IM and 0.9 x 10^8 PFU of MVA.tHIVconsv4 (M4) are administered IM simultaneously, one into the deltoid muscle of each arm.
  Interventions: Biological: Vaccine
- 2. Placebo (Placebo Comparator): Normal sterile saline (0.9% Sodium Chloride solution) administered IM as Placebo, the volume is matched to that of the vaccines and administered in the deltoid muscle of each arm at Week 0 and at week 4 .
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Vaccine — IM vaccination with ChAdOx1.tHIVconsv1, MVA.tHIVconsv3 and MVA.tHIVconsv4
  Arms: 1: Vaccine
Biological: Placebo — IM administration of 0.9% sterile sodium chloride solution
  Arms: 2. Placebo

SUMMARY:
HIV-CORE 006 is a Phase 1 double-blind placebo-controlled trial, in which the mosaic immunogens are delivered by a prime-boost regimen of non-replicating simian adenovirus followed by non-replicating poxvirus MVA. Volunteers will be randomised to receive either the vaccine regimen or placebo at 2 vaccination visits 4 weeks apart. The vaccine regimen consists of a single mosaic prime ChAdOx1.tHIVconsv1 (C1) and a dual boost of MVA.tHIVconsv3 (M3) and MVA.tHIVconsv4 (M4) administered simultaneously. The trial will recruit healthy African adults 18-50 years of age, who are HIV-uninfected and at low risk of HIV infection.

The trial is designed to enrol 88 healthy men and women, who will be randomised to receive either the vaccine regimen or placebo in a ratio of 72:16:

* Vaccine Arm (ChAdOx1.tHIVconsv1 prime followed by MVA.tHIVconsv3 and MVA.tHIVconsv4 boost at 4 weeks after enrolment); 72 vaccine recipients;
* Placebo Arm; 16 recipients

To maintain blinding, all volunteers will receive two injections with half dose into the deltoid region of each arm of ChAdOx1.tHIVconsv1 or placebo at enrolment, and two injections (MVA.tHIVconsv3 or placebo into one deltoid region and MVA.tHIVconsv4 or placebo into the other) at 4 weeks after enrolment. The primary goal of assessing safety and immunogenicity will be served by weighting the randomisation toward vaccinees.

DETAILED DESCRIPTION:
Phase 1 clinical trial HIV-CORE (COnserved REgions) 006 is a trial of a new combined vaccine regimen to determine safety and immunogenicity in healthy adults in Kenya, Uganda and Zambia. Immune responses may vary between populations and so it is important to confirm that the vaccines are suitable for the people and environment where they will be deployed for protection against HIV/AIDS. There are many different strains of HIV-1, and the virus can change to escape immune responses. This vaccine regimen is designed to work in all parts of the world.

The aim is to induce effective cytotoxic T lymphocytes (CTL) against HIV-1. These could complement broadly neutralizing antibodies in prophylaxis and play a central role in cure. CTL exert their effector functions by killing HIV-1-infected cells and producing soluble factors, which directly or indirectly counteract the HIV-1 replicative cycle. In future, this approach could be combined, in human efficacy testing, with other immunogens that stimulate humoral responses, with the goal of effectively preventing HIV-1 infections.

The central principle of this strategy is to focus T-cell immune responses on the most conserved regions of the HIV-1 proteome. These regions are common to most variants and, if mutated, reduce the ability of the virus to grow; these regions are the "Achilles heel" of HIV-1. Targeting of conserved regions is further enhanced by using 'mosaic' proteins, which are designed by computer to maximize the match of the vaccine with global HIV-1 variants and to block common ways the HIV-1 changes to escape the immune response. Vaccines should match circulating HIV-1 variants as much as possible to stop them efficiently. When T cells attack conserved parts of HIV-1 proteins (parts that seldom or never change), the disease is better controlled-this vaccine includes those parts.

The HIV-1-derived mosaic genes are called tHIVconsvX and are delivered by two safe, non-replicating vaccine vectors derived from chimpanzee adenovirus and poxvirus modified vaccinia virus Ankara (MVA). Adenoviruses, if able to grow, normally cause respiratory and gastrointestinal ailments, while the unmodified chimpanzee adenovirus is not known to cause disease in humans; the engineered vaccine vector called ChAdOx1 is crippled so it cannot grow. ChAdOx1 and similar experimental vaccines have been shown to be safe in over 1,500 human volunteers. MVA is a poxvirus, which does not replicate in humans. It was used safely as the smallpox vaccine in over 120,000 people at the end of the smallpox-eradication campaign and as an experimental vaccine vector against a variety of diseases in many clinical trials.

Humans and microbiota, which consist of bacteria, fungi, viruses and eukaryotic species, have co-evolved over millions of years and their coexistence is beneficial to both parties. Human immune system is constitutively exposed to microbial stimulation and any vaccine design and responsiveness needs to be considered in the context of host-microbiota interactions. Manipulation of the microbiota functions and composition through diet, engraftment and/or any other means may thus become a viable strategy for improving vaccine responsiveness as well as treating malfunctions of the immune system. The first reports on the influence of gut microbiota diversity and composition on responses to vaccination have been emerging for some time. As part of the exploratory endpoints for this trial, the gut microbiome of study volunteers will be characterised for composition and richness before and after administration of the study vaccines.

The ChAdOx1-vectored HIV-1 vaccine in this trial will be tested for the first time in humans, and MVA.tHIVconsv3 and MVA.tHIVconsv4 (M3M4) are currently administered to HIV-positive individuals in the first-in-human clinical trial in the USA (NCT03844386). However, this is the first time these C1-M3M4 vaccines will be administered to humans sequentially. In parallel with HIV-CORE 006, these vaccines will be tested for safety in the United Kingdom, in a phase I trial HIV-CORE 0052. The tHIVconsvX vaccines have been designed for global use irrespective of the HIV-1 strain and are therefore very suitable for Africa, where multiple strains are responsible for the epidemic, mainly from the HIV-1 families A, D and C. The HIV-CORE 006 trial will take place at four sites in Africa and will enrol healthy adults between 18 and 50 years of age. It is not yet known whether the vaccine will have a beneficial effect, no effect, or whether it could cause harm. The health of trial volunteers will be monitored carefully, and volunteers will receive counselling and support to minimise HIV-1 infection.

This trial is funded by EDCTP, under the SRIA-2015-1066 grant

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female as assessed by a medical history, physical exam, and laboratory tests.
* At low risk of HIV infection and willing to maintain low-risk behaviour for the duration of the trial. Individuals from key populations are not excluded provided they are assessed to be at low risk of HIV infection at screening and are willing to maintain low-risk behaviour during the study.
* At least 18 years of age on the day of screening and have not reached their 51st birthday on the day of the first vaccination.
* Willing and able to give informed consent for participation in the trial before any study-related procedures are performed. Volunteers will pass an Assessment of Understanding before signing the consent form.
* Willing to comply with the requirements of the protocol and be available for follow up for the planned duration of the study.
* Willing to undergo HIV testing, risk reduction counselling, receive HIV test results
* All sexually active males (unless anatomically sterile or in a monogamous relationship with a female partner who uses a documented non-barrier method of birth control) must be willing to use an effective method of contraception (such as consistent condom use) from the day of first vaccination until 4 months after the last vaccination.
* If a female of childbearing potential, willing to use an effective non-barrier method of contraception (hormonal contraceptive or intrauterine device) from at least 2 weeks prior to first vaccination until at least 4 months after the last study vaccination. If not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/L) or surgically sterile: no additional contraception required.
* All female volunteers must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures and must test negative prior to each study vaccination.
* Willing to forego donations of blood or any other tissues during the trial and, for those who test positive for HIV antibodies due to vaccination (vaccine-induced seropositivity/ reactivity), until the anti-HIV antibody titres become undetectable.

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection
* Receipt of any vaccine in the previous 28 days or planned receipt within 28 days of Investigational Medicinal Product. Volunteers who expect to receive any adenoviral vectored vaccines within the next three months after ChAdOx1.tHIVconsv1 vaccine administration should not participate due to the risk of immune interference with the study vaccine.
* Participation in another clinical trial of an Investigational Medicinal Product (IMP) currently, within the previous 3 months or expected participation during the study.
* Receipt of another investigational HIV vaccine candidate or investigational adenoviral vectored vaccine (Note: receipt of an HIV vaccine placebo will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval).
* Receipt of blood transfusion or blood-derived products within the previous 4 months or expectation of receiving blood products during the study period.
* Receipt of immunoglobulin products within the previous 3 months.
* If female, pregnant or planning a pregnancy during the period of enrolment until 4 months after the last study vaccination; or lactating.
* Any clinically relevant abnormality on history or examination such as:

  * Any confirmed or suspected history of immunodeficiency including recurrent severe infections;
  * Use of systemic corticosteroids for >14 days (use of topical or inhaled steroids is permitted) within the previous 6 months;
  * Immunosuppressive, anti-cancer, anti-tuberculosis or other medications considered significant by the investigator within the previous 6 months.
  * History of splenectomy.
  * History of autoimmune disease
  * Bleeding disorder diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions). (Note: a volunteer that states that he or she has easy bruising or bleeding but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience is eligible)
  * History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, or clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow up).
  * History of cancer (except basal cell carcinoma of the skin)
  * Asthma that is not well controlled.
  * History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
  * History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulty, angioedema).
  * History of Guillain-Barre syndrome.
  * Confirmed diagnosis of active or chronic hepatitis B, hepatitis C, active syphilis and/or active tuberculosis
  * Seizure disorder: an individual who has had a seizure in the last 3 years is excluded (Not excluded: an individual with a history of seizures who has neither required medication nor had a seizure for three or more years).
  * History of serious psychiatric conditions or any psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
  * Substance abuse disorder that precludes compliance with the protocol as assessed by the investigator.
  * Any clinically significant acute or chronic medical condition that is considered unstable/progressive, or in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Abnormal clinically significant abnormal finding on screening biochemistry or haematology blood, or urinalysis, including but not limited to:

Haematology:

* Haemoglobin - <9.5 g/dl in females; <11.0 g/dl in males
* Absolute Neutrophil Count (ANC) - ≤1,000/mm3
* Absolute Lymphocyte Count (ALC) - ≤650/mm3
* Platelets - <100,000 cells/mm3 Chemistry
* Creatinine >1.1 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) >1.25 x ULN
* Alanine aminotransferase (ALT) >1.25 x ULN Urinalysis

Clinically significant abnormal dipstick confirmed by microscopy:

* Protein = 2+ or more
* Blood = 2+ or more (not due to menses)
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the study
* If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Safety- local and systemic reactogenicity post vaccination | 7 days
  Proportion of volunteers with local and systemic reactogenicity events from Day 0 to Day 7 post vaccination
Safety - unsolicited Grade 3 or Grade 4 adverse events post vaccination | 28 days
  Proportion of volunteers with Grade 3 or 4 unsolicited adverse events through 28 days post final vaccination
Safety - vaccine related SAEs | 48 weeks
  Proportion of volunteers with vaccine related serious adverse events (SAEs) collected throughout the study period
Immunogenicity - HIV-1 specific T-cell responses | 44 weeks
  Proportion of vaccine recipients developing HIV-1-specific T-cell responses

SECONDARY OUTCOMES:
Immunogenicity- Analysis of T-cell responses | 44 weeks
  Frequency, breadth and duration of T-cell responses to conserved epitopes measured by interferon-gamma ELISPOT assay in each vaccine recipient
Immunogenicity- Inhibition of HIV-1 viruses | 44 weeks
  Breadth of inhibition of HIV-1 viruses representative of circulating viruses in Kenya, Uganda and Zambia and other global clades in the in vitro Virus Inhibition Assay

CONTACTS AND LOCATIONS:
Overall Officials: Walter Jaoko, MD, Principal Investigator — University of Nairobi; Pontiano Kaleebu, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; William Kilembe, MD, Principal Investigator — Center for Family Health Research in Zambia; Eduard Sanders, MD, Principal Investigator — KEMRI-Wellcome Trust; Paola Cicconi, MD, Principal Investigator — University of Oxford
Locations (4):
- Kenya (2):
  - Kenya Medical Research Institute Wellcome Trust Programme, Kilifi
  - Kenya AIDS Vaccine Institute for Clinical Research, Nairobi
- Medical Research and Uganda Virus Research Institute and London School of Hygiene & Tropical Medicine Uganda Research Unit, Masaka, Uganda
- Center for Family Health Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Study information will be made available through an open repository. The information to be made available will be anonymized so that there is no link to participants and will include data on safety, immune responses and any other data generated from samples obtained in this study.
Supporting Information: Study Protocol
Time Frame: Within 12 months of the study completion date we will provide the additional document types as described above.
Access Criteria: Aim is to provide a summary of the results or a link to summary results within the trial registration record.

REFERENCES:
- [Derived] Chanda C, Kibengo F, Mutua M, Ogada F, Muturi-Kioi V, Akis Yildirim BM, Amondi M, Baines A, Basajja V, Borthwick N, Bosire K, Chambula E, Chetty P, Chinyenze K, Chirro O, Crook A, De Bont J, Fernandez N, Ejou P, Farah B, Glaze M, Gombe B, Gumbe A, Hayes P, Itwi S, Juma S, Kabarambi A, Kabengele C, Kafeero P, Kakande A, Kanungi J, Kidega W, King D, Mahira R, Malogo R, Matsoso M, Michelo C, Moyo A, Mugaba S, Mugenya I, Muhumuza P, Mujadidi YF, Muriuki M, Musale V, Mutua G, Muwowo M, Mwale F, Mwangi I, Nakimbugwe M, Namuyanja A, Nduati E, Nielsen L, Nyange J, Oino G, Okech B, Omosa-Manyonyi G, Otieno D, Palmer S, Phiri H, Ramko K, Rutishauser RL, Sayeed E, Sajabi R, Serwanga J, G-T Wee E, Wenden C, Cicconi P, Fast P, Gilmour J, Jaoko W, Kaleebu P, Kilembe W, Kuipers H, Sanders EJ, Hanke T. Safety and broad immunogenicity of HIVconsvX conserved mosaic candidate T-cell vaccines vectored by ChAdOx1 and MVA in HIV-CORE 006: a double-blind, randomised, placebo-controlled phase 1 trial in healthy adults living without HIV-1 in eastern and southern Africa. Lancet Microbe. 2025 Jun;6(6):101041. doi: 10.1016/j.lanmic.2024.101041. Epub 2025 May 16. PMID 40388952